CLINICAL TRIAL: NCT00798629
Title: A Dose Ranging Trial of Adenovirus CCL-21 Transduced MART-1/gp100 Peptide-Pulsed Dendritic Cells Matured Using Cytokines for Patients With Chemotherapy-Resistant Metastatic Melanoma
Brief Title: Adenovirus CCL-21 Transduced MART-1/gp100/Tyrosinase/NY-ESO-1 Peptide-Pulsed Dendritic Cells Matured
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15280; NCI P-8190 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma; mucosal melanoma
MeSH Terms: conditions — Melanoma | interventions — Peptides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vaccine Dose Escalation (Experimental): Dose Escalation: Intradermal DC Injection. Level 1: Cell Dose: 2 x 10^6 Level 2: Cell Dose: 1 x 10^7 Level 3: Cell Dose: 2 x 10^7
  Interventions: Biological: Autologous dendritic cell-adenovirus CCL21 vaccine

INTERVENTIONS:
Biological: Autologous dendritic cell-adenovirus CCL21 vaccine — Intradermal injections of adenovirus-CCL-21 transduced class I peptide-pulsed DC
  Other Names: gp100:209-217(210M)Peptide; NSC 683472; MART-1:26-35(27L)Peptide; NSC 709401; dendritic cell (DC)

SUMMARY:
RATIONALE: Vaccines made from gene-modified tumor cells may help the body build an immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
In this phase I study, patients will receive intradermal injections of adenovirus-CCL-21 transduced class I peptide-pulsed DC with total volumes for each intradermal injection of no more than 1 ml to be split into four injections of 0.25 ml each in four limbs in node draining areas (proximal arms and thighs), for a total DC dose of 2 X 10^6, 10^7 or 2 X 10^7 cells to be administered intradermally. DC injections in one course of therapy will be given four times at intervals of weekly for two doses (days 1 and 8 +/- 72 hrs.), then every two weeks for two doses (at days 22 +/- 72 hrs. and 36 +/- 72 hours). Cells will be harvested for DC administration and a flow cytometry analysis as well as microbiologic analysis including bacterial/fungal cultures and gram stain will be performed prior to infusion. All injections will be based on number of DC, not number of total cells.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic melanoma with measurable disease after attempted curative surgical therapy and who have received at least one prior chemotherapy regimen; adjuvant interferon or isolated limb perfusion is allowed.
* Tumor tissue must be available for immunohistochemical analysis, and specimens will stained for MART-1 by immunohistochemical staining and will also be stained for HMB-45 by immunohistochemistry, and positivity for at least one will be an entry requirement.
* Patients must be HLA-A *0201 positive, by a DNA SSOP analysis.
* Serum creatinine of 2.0 mg/dl or less, total bilirubin of 2.0 mg/dl or less, and ALT/AST of less than 3X institutional upper limit of normal.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients must be able to understand and sign an IRB approved informed consent form.
* Patients must have white blood count of 3000 or greater, platelets of 100,000 or greater, and hemoglobin of 9.0 gm/dl or more.
* Patients with unresectable stages III/IV uveal melanoma and metastatic mucosal melanoma will be eligible for this trial.

Exclusion Criteria:

* Undergoing or have undergone in the past month any other therapy for their melanoma, including radiation therapy, chemotherapy and adjuvant therapy
* Have major systemic infections, coagulation disorders, or other major medical illnesses of the cardiovascular or respiratory systems, or have had a documented MI in the last 6 months
* Require steroid therapy
* Patients who are pregnant or lactating
* Known to be positive for hepatitis BsAg, Hepatitis C or HIV antibody
* Have a prior history of uveitis or autoimmune inflammatory eye disease
* Have had another malignancy other than cervical carcinoma-in-situ or basal cell /squamous cancer of the skin, unless they have undergone curative therapy more than 3 years ago and are still free of detectable disease, since the effects of peptide-pulsed DC on other active cancers are unknown

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Immune response | 2 years, 5 months
  Assessment of immune responses to the cytokine-cocktail-matured class I peptide-pulsed adenoviral CCL-21 transduced DC cell vaccine. Immune reactivity will be monitored for the appearance of lymphoid-like structures at the vaccine site (as a result of CCL-21 production), in the blood for MART-1 /gp100 specific T cell frequency by tetramer based flow cytometry and ELISPOT analysis of fresh cells, and CTL cytolytic reactivity after in vitro sensitization prior to, four weeks after, and 8 weeks after immunization.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 2 years, 5 months
  Toxicity as assessed by NCI CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Weber, MD, PhD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States